CLINICAL TRIAL: NCT02639936
Title: Performance of a New Generation IGRA in Immunocompromised Individuals
Brief Title: New Generation IGRA in Immunocompromised Individuals
Acronym: TBnet#54
Status: Completed | Type: Observational
Sponsor: Tuberculosis Network European Trialsgroup (Network)
Responsible Party: Principal Investigator, Martina Sester, PhD, Head of Department, Tuberculosis Network European Trialsgroup
Other Study IDs: TBnet study #54
Record Dates: First submitted 2015-12-15; First posted 2015-12-28 (Estimated); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Monitoring, Immunologic; Active Tuberculosis; Tuberculosis in Solid Organ Transplant Recipients; Tuberculosis in Marrow Transplant Recipients; Tuberculosis in Rheumatoid Arthritis; Tuberculosis in Chronic Renal Failure; Tuberculosis in HIV-infected Individuals
MeSH Terms: conditions — Latent Tuberculosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Stimulated plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Immunocompetent controls: Control persons without immunodeficiency with and without active tuberculosis, with and without risk factors for prior exposure with M. tuberculosis
- Solid organ transplant recipients: Patients after solid organ transplantation with and without active tuberculosis, with and without risk factors for prior exposure with M. tuberculosis
- Stem cell transplant recipients: Patients after stem cell transplantation with and without active tuberculosis, with and without risk factors for prior exposure with M. tuberculosis
- Patients with rheumatoid arthritis: Patients with rheumatoid arthritis with and without active tuberculosis, with and without risk factors for prior exposure with M. tuberculosis
- Patients with chronic renal failure: Patients with chronic renal failure with and without active tuberculosis, with and without risk factors for prior exposure with M. tuberculosis
- Individuals with HIV infection: Individuals with HIV infection with and without active tuberculosis, with and without risk factors for prior exposure with M. tuberculosis

SUMMARY:
Evaluation of a new ELISA based interferon-gamma release assay (QuantiFERON TB plus In-tube test) in immunocompromized patients

DETAILED DESCRIPTION:
This study is designed to evaluate the performance of a new ELISA based QuantiFERON-TB plus In-tube test to identify M. tuberculosis specific immune Responses as evidence of latent infection with M. tuberculosis in immunosuppressed populations. Both qualitative and quantitative test results will be related to the level of immunodeficiency and to the presence of risk factors for prior exposure with M. tuberculosis. In addition, patients with active tuberculosis (both immunocompetent and immunocompromised individuals) will be included to evaluate a potential increase in sensitivity in these groups. Immunocompetent individuals with low risk of exposure will be analysed as a proxy to estimate specificity. Finally, this study will be extended to longitudinally assess the predictive value of a positive blood test for progression to active disease.

ELIGIBILITY:
Inclusion Criteria:

* Individuals as specified for the study Population
* Written informed consent

Exclusion Criteria:

* <18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Immunocompetent and immunocompromised patients
Sampling Method: Non-Probability Sample
Enrollment: 2663 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2023-12 (Actual); Study Completion 2023-12 (Actual)

PRIMARY OUTCOMES:
Specificity | 2 years
  The percentage of negative test results will be quantified among controls and patients without risk factors for M. tuberculosis exposure.
Sensitivity | 2 years
  The percentage of positive test results will be quantified among controls and patients with active tuberculosis.
Indeterminate results | 2 years
  The percentage of indeterminate results will be quantified in immunocompetent and immunocompromised patients
Association with exposure | 2 years
  Results from QFT-Plus assay will be associated with risk factors for M. tuberculosis exposure
Progression | 4 years
  The number of individuals progressing to tuberculosis will be quantified depending on the test result at the time of screening and depending on preventive chemotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Martina Sester, PhD, Principal Investigator — Universität des Saarlandes
Locations (16):
- Rigshospitalet, Copenhagen, Denmark
- Germany (3):
  - Research center Borstel, Borstel
  - Freiburg University, Freiburg im Breisgau
  - Saarland University, Homburg
- Italy (3):
  - University of Brescia and Brescia Spedali Civili General Hospital, Brescia
  - San Raffaele Scientific institute, Milan
  - National Institute for Infectious Diseases L. Spallanzani, Rome
- Department of Pneumology & Allergology, Chisinau, Moldova
- Department of Infectious Diseases; Oslo University, Oslo, Norway
- Warszawski Uniwersytet Medyczny, Warsaw, Poland
- Centro de Diagnóstico Pneumológico, Vila Nova de Gaia, Portugal
- Marius Nasta Institute of Pneumology, Bucharest, Sector 5, Romania
- Spain (3):
  - Institut d'Investigació Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Central de Asturias, Oviedo
- Department of Respiratory Medicine, Royal Free Hospital, London, United Kingdom

REFERENCES:
- [Derived] Sester M, Altet-Gomez N, Andersen AB, Arias-Guillen M, Avsar K, Bakken Kran AM, Bothamley G, Nordholm Breschel AC, Brown J, Chesov D, Ciobanu N, Cirillo DM, Crudu V, de Souza Galvao M, Dilektasli AG, Dominguez J, Duarte R, Dyrhol-Riise AM, Goletti D, Hoffmann H, Ibraim E, Kalsdorf B, Krawczyk M, Kunst H, Lange B, Lipman M, Matteelli A, Milkiewicz P, Neyer D, Nitschke M, Oral HB, Palacios-Gutierrez JJ, Petruccioli E, Raszeja-Wyszomirska J, Ravn P, Rupp J, Spohn HE, Toader C, Villar-Hernandez R, Wagner D, van Leth F, Martinez L, Pedersen OS, Lange C. Diagnostic accuracy and predictive value of the QuantiFERON-TB gold plus assay for tuberculosis in immunocompromised individuals: a prospective TBnet study. Lancet Reg Health Eur. 2025 Aug 6;57:101416. doi: 10.1016/j.lanepe.2025.101416. eCollection 2025 Oct. PMID 40823191
- See also: TBnet website — http://www.tb-net.org